CLINICAL TRIAL: NCT01414608
Title: A Phase III Trial of Adjuvant Chemotherapy Following Chemoradiation as Primary Treatment for Locally Advanced Cervical Cancer Compared to Chemoradiation Alone: The OUTBACK Trial
Brief Title: Cisplatin and Radiation Therapy With or Without Carboplatin and Paclitaxel in Patients With Locally Advanced Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZGOG-0902-GOG-0274; NCI-2011-02978 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANZGOG-0902/GOG-0274/RTOG-1174; CDR0000706698; GOG-0274; RTOG-1174; ANZGOG-0902; S12-01864; ANZGOG-0902-GOG-0274 (Other: NRG Oncology); ANZGOG-0902-GOG-0274 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Stage IB Cervical Cancer AJCC v6 and v7; Stage IIA Cervical Cancer AJCC v7; Stage IIB Cervical Cancer AJCC v6 and v7; Stage IIIB Cervical Cancer AJCC v6 and v7; Stage IVA Cervical Cancer AJCC v6 and v7
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiation; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cisplatin, radiation therapy, brachytherapy) (Experimental): Patients receive cisplatin IV over 60-90 minutes on days 1, 8, 15, 22, and 29. Patients also undergo external-beam radiation therapy once daily, 5 days a week, for approximately 5 weeks. Patients then undergo high-dose rate, pulsed-dose rate, or low-dose rate intracavitary brachytherapy.
  Interventions: Radiation: Brachytherapy; Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Other: Quality-of-Life Assessment
- Arm II (cisplatin, radiation therapy, brachytherapy, chemo) (Experimental): Patients receive cisplatin and undergo external-beam radiation and brachytherapy as in arm I. Beginning 4 weeks later, patients also receive adjuvant chemotherapy comprising paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Brachytherapy; Drug: Carboplatin; Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Radiation: Brachytherapy — Undergo brachytherapy
  Other Names: Brachytherapy, NOS; Internal Radiation; Internal Radiation Brachytherapy; Internal Radiation Therapy; Radiation Brachytherapy; Radiation, Internal
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm II (cisplatin, radiation therapy, brachytherapy, chemo)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm II (cisplatin, radiation therapy, brachytherapy, chemo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies how well giving cisplatin and radiation therapy together with or without carboplatin and paclitaxel works in treating patients with cervical cancer has spread from where it started to nearby tissue or lymph nodes. Drugs used in chemotherapy, such as cisplatin, carboplatin, and paclitaxel, work in different ways to stop the growth of [cancer/tumor] cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. External radiation therapy uses high-energy x rays to kill tumor cells. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. It is not yet known whether giving cisplatin and external and internal radiation therapy together with carboplatin and paclitaxel kills more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the addition of adjuvant chemotherapy to standard cisplatin-based chemoradiation improves overall survival.

SECONDARY OBJECTIVES:

I. To determine the progression-free survival rates. II. To determine acute and long-term toxicities. III. To determine patterns of disease recurrence. IV. To determine the association between radiation protocol compliance and outcomes.

V. To determine patient quality of life, including psycho-sexual health.

TERTIARY OBJECTIVES:

I. To determine the association between the results of a follow-up positron emission tomography (PET) scan performed 4-6 months post completion of chemoradiation and outcomes for all patients in the trial.

II. To determine the biological predictors of patients' outcomes based on translational laboratory studies of blood and tissue specimens.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cisplatin intravenously (IV) over 60-90 minutes on days 1, 8, 15, 22, and 29. Patients also undergo external-beam radiation therapy once daily, 5 days a week, for approximately 5 weeks. Patients then undergo high-dose rate, pulsed-dose rate, or low-dose rate intracavitary brachytherapy.

ARM II: Patients receive cisplatin and undergo external-beam radiation and brachytherapy as in arm I. Beginning 4 weeks later, patients also receive adjuvant chemotherapy comprising paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients may undergo baseline tumor biopsy and blood collection for future correlative studies.

Patients complete the European Organization for Research and Treatment of Cancer (EORTC) Core questionnaire (QLQ-C30), the EORTC cervix cancer module (CX24), the ovarian cancer module (OV28), and the Sexual function-Vaginal Changes Questionnaire (SVQ) questionnaires at baseline, during, and after completion of study treatment.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will have locally advanced cervical cancer suitable for primary treatment with chemoradiation with curative intent, in addition to:

  * Federation of Gynecology and Obstetrics (FIGO) 2008 stage IB1 & node positive, IB2, IIA, IIB, IIIB, or IVA disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Histological diagnosis of squamous cell carcinoma, adenocarcinoma or adenosquamous cell carcinoma of the cervix
* White blood cells (WBC) >= 3.0 x 10^9/L
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 x ULN (if both tests are done, both results need to be =< 2.5 x ULN)
* Creatinine =< ULN (Common Toxicity Criteria [CTC] grade 0) OR calculated creatinine clearance (Cockcroft-Gault formula) >= 60 mL/min OR >= 50 mL/min by ethylenediaminetetraacetic acid (EDTA) creatinine clearance
* Written informed consent

Exclusion Criteria:

* Any previous pelvic radiotherapy
* Para-aortic nodal involvement above the level of the common iliac nodes or L3/L4 (if biopsy proven, PET positive, or >= 15 mm short-axis diameter on computed tomography [CT])
* FIGO 2008 stage IIIA disease
* Patients assessed at presentation as requiring interstitial brachytherapy treatment
* Patients with bilateral hydronephrosis unless at least one side has been stented and renal function fulfills the required inclusion criteria
* Previous chemotherapy for this tumor
* Evidence of distant metastases
* Prior diagnosis of Crohn's disease or ulcerative colitis
* Peripheral neuropathy >= grade 2 (per Common Terminology Criteria for Adverse Events [CTCAE] version [v]4)
* Patients who have undergone a previous hysterectomy or will have a hysterectomy as part of their initial cervical cancer therapy; this includes patients with a prior history of supracervical hysterectomy
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer and in situ melanoma, who had (or have) any evidence of the other cancer present within the last 5 years
* Patients who are pregnant or lactating
* Any contraindication to the use of cisplatin, carboplatin, or paclitaxel chemotherapy
* Serious illness or medical condition that precludes the safe administration of the trial treatment including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are known to be human immunodeficiency virus (HIV) positive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 926 (Actual)
Dates: Start 2012-01-09 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen N Moore, Principal Investigator — NRG Oncology
Locations (326):
- United States (315):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Oncology Associates-Biltmore Cancer Center, Phoenix, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - Arizona Oncology Associates-Wilmot, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - New York Hospital Medical Center of Queens, Fresh Meadows, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Queens Hospital Center, Jamaica, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Toledo, Toledo, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Texas Oncology at Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (8):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Zhongshan Hospital Fudan University, Guangdong Province, Shanghai Municipality, China
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia
- National University Hospital Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Mileshkin LR, Moore KN, Barnes EH, Gebski V, Narayan K, King MT, Bradshaw N, Lee YC, Diamante K, Fyles AW, Small W Jr, Gaffney DK, Khaw P, Brooks S, Thompson JS, Huh WK, Mathews CA, Buck M, Suder A, Lad TE, Barani IJ, Holschneider CH, Van Dyk S, Quinn M, Rischin D, Monk BJ, Stockler MR. Adjuvant chemotherapy following chemoradiotherapy as primary treatment for locally advanced cervical cancer versus chemoradiotherapy alone (OUTBACK): an international, open-label, randomised, phase 3 trial. Lancet Oncol. 2023 May;24(5):468-482. doi: 10.1016/S1470-2045(23)00147-X. Epub 2023 Apr 17. PMID 37080223
- [Derived] Gould HJ 3rd, Miller PR, Edenfield S, Sherman KJ, Brady CK, Paul D. Emergency Use of Targeted Osmotic Lysis for the Treatment of a Patient with Aggressive Late-Stage Squamous Cell Carcinoma of the Cervix. Curr Oncol. 2021 Jun 8;28(3):2115-2122. doi: 10.3390/curroncol28030196. PMID 34201380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open to accrual on January 9th 2012. Accrual ended on June 28th 2017
Groups:
- Standard Chemoradiation: Standard Chemoradiation (CRT)
- Standard Chemoradiation With Adjuvant Chemotherapy: Standard Chemoradiation (CRT) followed by 4 cycles of carboplatin and paclitaxel (Adjuvant)
Period: Overall Study
Arm/Group | Standard Chemoradiation | Standard Chemoradiation With Adjuvant Chemotherapy
Started | 461 | 465
Completed | 456 | 463
Not Completed | 5 | 2
Not completed — Ineligible | 5 | 2

BASELINE CHARACTERISTICS:
Population: Eligible subjects
Groups:
- Standard Chemoradiation: patients receive 45 - 50.4 Gy external beam radiation therapy (EBRT) delivered in fractions of 1.8 Gy to the pelvis, followed by brachytherapy. Cisplatin was given during the radiation at a dose of 40mg/m2 weekly for 5 doses to all patients.
- Standard Chemoradiation With Adjuvant Chemotherapy: patients receive 45 - 50.4 Gy external beam radiation therapy (EBRT) delivered in fractions of 1.8 Gy to the pelvis, followed by brachytherapy. Cisplatin will be given during the radiation at a dose of 40mg/m2 weekly for 5 doses to all patients. Within 4 weeks of completion of all radiation treatment, and following recovery from toxicities, patients in Arm B were treated with an additional 4 cycles of 3 weekly adjuvant chemotherapy using carboplatin AUC 5 and paclitaxel 155 mg/m2.
- Total: Total of all reporting groups
Arm/Group | Standard Chemoradiation | Standard Chemoradiation With Adjuvant Chemotherapy | Total
Number analyzed (Participants) | 456 | 463 | 919
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 139 | 146 | 285
  40 - 49 years | 148 | 130 | 278
  50 - 59 years | 103 | 117 | 220
  > 60 years | 66 | 70 | 136
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 456 | 463 | 919
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The American Indian group also includes Aboriginal/Torres Strait Islander/Native American. The Australian study developers report race using this group rather than American Indian
  Participants
    American Indian or Alaska Native | 7 | 7 | 14
    Asian | 22 | 31 | 53
    Native Hawaiian or Other Pacific Islander | 4 | 6 | 10
    Black or African American | 68 | 53 | 121
    White | 326 | 337 | 663
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate at 5 Years
Description: Estimate for probability of overall survival at 5 years by Kaplan-Meier method, where overall survival is defined as the time from randomization to time of death due to any cause or the date of last contact, whichever occurs first.
Time Frame: 5 years from study randomization
Population: Eligible subjects
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Standard Chemoradiation: Patients receive 45 - 50.4 Gy external beam radiation therapy (EBRT) delivered in fractions of 1.8 Gy to the pelvis, followed by brachytherapy. Cisplatin given during the radiation at a dose of 40mg/m2 weekly for 5 doses
- Standard Chemoradiation With Adjuvant Chemotherapy: patients receive 45 - 50.4 Gy external beam radiation therapy (EBRT) delivered in fractions of 1.8 Gy to the pelvis, followed by brachytherapy. Cisplatin given during the radiation at a dose of 40mg/m2 weekly for 5 doses. Within 4 weeks of completion of all radiation treatment, and following recovery from toxicities, patients were treated with an additional 4 cycles of 3 weekly adjuvant chemotherapy using carboplatin AUC 5 and paclitaxel 155 mg/m2.
Arm/Group | Standard Chemoradiation | Standard Chemoradiation With Adjuvant Chemotherapy
Number analyzed (Participants) | 456 | 463
Percentage of participants | 71 [66 to 75] | 72 [67 to 76]

2. Secondary Outcome: Progression-free Survival Rate at 5 Years
Description: Estimate for probability of progression free at 5 years by Kaplan-Meier method, where progression-free survival is defined as the time from randomization to the time of disease progression, death from any cause or date of last contact, whichever occurs first. Disease progression is defined by increasing clinical, radiological or pathological evidence of disease from participant entry to when investigator deems a progression. RECIST V1.0 was not used to determine response on this study.
Time Frame: 5 years from study randomization
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard Chemoradiation | Standard Chemoradiation With Adjuvant Chemotherapy
Number analyzed (Participants) | 456 | 463
Percentage of participants | 62 [57 to 66] | 63 [58 to 68]

3. Secondary Outcome: Number of Participants With Adverse Events (Grade 3 or Higher) in First Year
Description: Number of participants with a maximum grade of 3 or higher for pre-specified adverse events that occurred during the first year after randomization. Adverse events are graded and categorized using CTCAE v4.0.
Time Frame: 1 year after randomization
Population: Arm A:eligible participants who received at least one dose of cisplatin and/or any dose of radiotherapy. Arm B: eligible participants who received at least one dose of adjuvant chemotherapy (carboplatin, paclitaxel, cisplatin or docetaxel)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Chemoradiation | Standard Chemoradiation With Adjuvant Chemotherapy
Number analyzed (Participants) | 453 | 361
Participants
  Abdominal pain | 13 | 14
  Alanine aminotransferase increased | 4 | 2
  Allergic reaction/hypersensitivity | 1 | 2
  Alopecia | 0 | 1
  Anemia | 32 | 64
  Aspartate aminotransferase increased | 3 | 2
  Colitis | 2 | 2
  Colonic obstruction | 1 | 1
  Creatinine Increased | 3 | 3
  Cystitis noninfective | 1 | 3
  Dehydration | 13 | 9
  Dermatitis radiation | 1 | 1
  Diarrhea | 21 | 20
  Enterocolitis | 2 | 3
  Fatigue | 7 | 9
  Febrile Neutropenia | 9 | 9
  Female genital tract fistula | 4 | 1
  Hearing impaired | 0 | 4
  Hemorrhage bladder | 3 | 3
  Hemorrhage rectum | 1 | 0
  Lymphocyte count decreased | 208 | 211
  Mucositis oral | 2 | 0
  Myalgia | 0 | 3
  Nausea | 11 | 11
  Neutrophil count decreased | 33 | 71
  Pain in extremity | 3 | 1
  Pelvic pain | 11 | 6
  Perineal pain | 1 | 0
  Peripheral motor neuropathy | 0 | 4
  Peripheral sensory neuropathy | 1 | 16
  Platelet count decreased | 5 | 16
  Proctitis | 2 | 0
  Small intestinal obstruction | 1 | 4
  Thrombosis/Thrombus/Embolism | 7 | 7
  Tumor pain | 6 | 0
  Urinary tract pain | 1 | 0
  Uterine obstruction | 1 | 2
  Vaginal Dryness | 0 | 1
  Vaginal pain | 3 | 1
  Vaginal stricture | 4 | 4
  Vomiting | 9 | 15

4. Secondary Outcome: Patterns of Disease Recurrence
Description: Number of patients for the site of disease recurrence. Disease was considered as persistent if participant had evidence of disease at study entry and disease did not progress during study. Disease status was considered locoregional alone if a participant had disease progression in the pelvis region including vagina after study entry. Disease status was considered distant if a participant had disease progression outside the pelvis (for example the abdomen and lung) after study entry. Criteria used to determine the no progression group includes participants that expired without documentation of progression.
Time Frame: through study completion an average of 60 months
Population: Eligible participants. The "No Progression recorded group" included participants who died due to any causes without documented progression.
Measure: Number; unit: participants
Arm/Group | Standard Chemoradiation | Standard Chemoradiation With Adjuvant Chemotherapy
Number analyzed (Participants) | 456 | 463
participants
  Persistent | 15 | 5
  Locoregional alone | 33 | 47
  Distant with or without locoregional | 51 | 42
  Other/Unknown | 53 | 37
  No Progression recorded | 304 | 332

5. Secondary Outcome: Radiation Protocol Compliance
Description: Radiation protocol compliance measured by external beam dose delivered
Time Frame: Average duration of 7 weeks
Population: Eligible and received radiotherapy
Measure: Mean (Full Range); unit: Gray
Groups:
- Arm A: Patients receive 45 - 50.4 Gy external beam radiation therapy (EBRT) delivered in fractions of 1.8 Gy to the pelvis, followed by brachytherapy. Cisplatin given during the radiation at a dose of 40mg/m2 weekly for 5 doses
- Arm B: patients receive 45 - 50.4 Gy external beam radiation therapy (EBRT) delivered in fractions of 1.8 Gy to the pelvis, followed by brachytherapy. Cisplatin given during the radiation at a dose of 40mg/m2 weekly for 5 doses. Within 4 weeks of completion of all radiation treatment, and following recovery from toxicities, patients were treated with an additional 4 cycles of 3 weekly adjuvant chemotherapy using carboplatin AUC 5 and paclitaxel 155 mg/m2.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 450 | 448
Gray | 45.6 [1.8 to 85.0] | 45.7 [4.5 to 90.0]

6. Secondary Outcome: Quality of Life for Global Health Status
Description: Quality of Life measured by change of global health status score from baseline to 12 months follow-up. A cancer-specific questionnaire with 30 items which summarize as five functioning scales, a global health status/quality of life scale, three symptom scales and six single items assessing additional symptoms and perceived financial impact. The minimum global health status score was 0 and the maximum global health status score was 100. A higher global health status score means better outcome.
Time Frame: Baseline and 12 months
Population: Eligible participants with Quality of Life at baseline and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Chemoradiation | Standard Chemoradiation With Adjuvant Chemotherapy
Number analyzed (Participants) | 165 | 174
score on a scale | 1.7 (22.8) | 2.4 (26.3)

ADVERSE EVENTS:
Time Frame: Through study completion with a median follow-up being 60 months.
Description: Specific Serious Adverse Events were not provided, an overall number was provided. Therefore, the term "General disorders" was used to satisfy reporting requirements. All-Cause Mortality includes all eligible participants. Serious Adverse Events and Other Adverse Events include only eligible participants who received at least one dose of cisplatin and/or any dose of radiotherapy for Standard Chemo arm and eligible participants who received at least one dose of adjuvant chemo in the second arm
Groups:
- Standard Chemoradiation: 45 - 50.4 Gy external beam radiation therapy (EBRT) delivered in fractions of 1.8 Gy to the pelvis, followed by brachytherapy. Cisplatin given during the radiation at a dose of 40mg/m2 weekly for 5 doses. At risk population includes eligible participants who received at least one dose of cisplatin and/or any dose of radiotherapy.
- Standard Chemoradiation With Adjuvant Chemotherapy: 45 - 50.4 Gy external beam radiation therapy (EBRT) delivered in fractions of 1.8 Gy to the pelvis, followed by brachytherapy. Cisplatin given during the radiation at a dose of 40mg/m2 weekly for 5 doses to all patients. Within 4 weeks of completion of all radiation treatment, and following recovery from toxicities, participants were treated with an additional 4 cycles of 3 weekly adjuvant chemotherapy using carboplatin AUC 5 and paclitaxel 155 mg/m2. At risk population includes eligible participants who received at least one dose of adjuvant chemotherapy (carboplatin, paclitaxel, cisplatin or docetaxel).
Arm/Group | Standard Chemoradiation | Standard Chemoradiation With Adjuvant Chemotherapy
All-Cause Mortality (participants affected / at risk) | 123/456 | 109/463
Serious Adverse Events (participants affected / at risk) | 98/453 | 107/361
Other Adverse Events (participants affected / at risk) | 438/453 | 360/361
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Chemoradiation (N=453) | Standard Chemoradiation With Adjuvant Chemotherapy (N=361)
General disorders NOS (General disorders) | 98 (98) | 107 (107) — Specific Adverse Events were not provided, an overall number was provided. Therefore, General disorder is used to satisfy reporting requirements.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Chemoradiation (N=453) | Standard Chemoradiation With Adjuvant Chemotherapy (N=361)
Abdominal pain (Gastrointestinal disorders) | 160 | 164
Alanine aminotransferase increased (Investigations) | 76 | 98
Allergic reaction/ hypersensitivity (Immune system disorders) | 20 | 32
Alopecia (Skin and subcutaneous tissue disorders) | 36 | 285
Anal pain (Gastrointestinal disorders) | 15 | 6
Anemia (Blood and lymphatic system disorders) | 293 | 303
Aspartate aminotransferase increased (Investigations) | 43 | 84
Colitis (Gastrointestinal disorders) | 12 | 16
Colonic obstruction (Gastrointestinal disorders) | 1 | 2
Creatinine increased (Investigations) | 53 | 58
Cystitis noninfective (Renal and urinary disorders) | 91 | 79
Dehydration (Metabolism and nutrition disorders) | 53 | 57
Dermatitis radiation (Injury, poisoning and procedural complications) | 65 | 65
Diarrhea (Gastrointestinal disorders) | 332 | 291
Enterocolitis (Gastrointestinal disorders) | 7 | 10
Fatigue (General disorders) | 358 | 333
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 9
Female genital tract fistula (Reproductive system and breast disorders) | 10 | 4
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 0 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 41 | 52
Hemorrhage Bladder (Renal and urinary disorders) | 44 | 43
Hemorrhage Rectum (Gastrointestinal disorders) | 31 | 35
Lymphedema (Vascular disorders) | 12 | 16
Lymphocyte count decreased (Investigations) | 320 | 287
Mucositis oral (Gastrointestinal disorders) | 27 | 37
Myalgia (Musculoskeletal and connective tissue disorders) | 44 | 142
Nausea (Gastrointestinal disorders) | 346 | 303
Neutrophil count decreased (Investigations) | 117 | 187
Pain in extremity (Musculoskeletal and connective tissue disorders) | 72 | 91
Pelvic pain (Reproductive system and breast disorders) | 128 | 110
Perineal pain (Reproductive system and breast disorders) | 8 | 4
Peripheral motor neuropathy (Nervous system disorders) | 10 | 68
Peripheral sensory neuropathy (Nervous system disorders) | 107 | 278
Platelet count decreased (Investigations) | 142 | 207
Proctitis (Gastrointestinal disorders) | 34 | 21
Rectal obstruction (Gastrointestinal disorders) | 1 | 0
Rectal pain (Gastrointestinal disorders) | 18 | 17
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 4
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 7 | 6
Thrombosis/Thrombus/Embolism (Hepatobiliary disorders) | 26 | 25
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 2
Urinary tract pain (Renal and urinary disorders) | 28 | 38
Uterine obstruction (Reproductive system and breast disorders) | 1 | 2
Vaginal discharge (Reproductive system and breast disorders) | 142 | 131
Vaginal dryness (Reproductive system and breast disorders) | 34 | 25
Vaginal pain (Reproductive system and breast disorders) | 50 | 34
Vaginal stricture (Reproductive system and breast disorders) | 31 | 14
Vomiting (Gastrointestinal disorders) | 165 | 174

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT01414608/Prot_SAP_ICF_000.pdf